CLINICAL TRIAL: NCT06316466
Title: Lipoprotein a is an Independent Risk Factor for Overall Survival in Patients With Pancreatic Cancer: a Propensity Score Matching Analysis
Status: Recruiting | Type: Observational
Sponsor: jingxue (Other)
Responsible Party: Sponsor-Investigator, jingxue, Associate professor, The Affiliated Hospital of Qingdao University
Organization: The Affiliated Hospital of Qingdao University (Other)
Other Study IDs: QYFYWZLL28521
Record Dates: First submitted 2024-03-12; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Pancreatic Carcinoma; Lipoprotein a; Overall Survival; Prognosis
Keywords: Pancreatic carcinoma; Lipoprotein a; Overall survival; Prognosis
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Apolipoproteins A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- the high Lp (a) groups and the low Lp (a) groups: The cut-off value for Lp (a) was determined based on one-year survival rates after diagnosis. Patients were then categorized into the high and low Lp (a) groups.
  Interventions: Other: Lp(a)
- the low Lp (a) groups: The cut-off value for Lp (a) was determined based on one-year survival rates after diagnosis. Patients were then categorized into the high and low Lp (a) groups.
  Interventions: Other: Lp(a)

INTERVENTIONS:
Other: Lp(a) — The cut-off value for Lp (a) was determined based on one-year survival rates after diagnosis. Patients were then categorized into the high and low Lp (a) groups.

SUMMARY:
Background: This study aims to assess the prognostic significance of serum lipoprotein (a) [Lp (a)] levels on overall survival (OS) and progression free survival (PFS) in individuals diagnosed with pancreatic cancer through the utilization of propensity score matching (PSM).

Methods: A retrospective analysis was conducted on the clinicopathological data of 364 patients diagnosed with pancreatic cancer at the Affiliated Hospital of Qingdao University from January 2019 to December 2022. The cut-off value for Lp (a) was determined based on one-year survival rates after diagnosis. Patients were then categorized into the high and low Lp (a) groups. We applied PSM analysis to minimize selection bias. The study compared OS and PFS between two groups by Kaplan-Meier method and analyzed differences using the log-rank test. Additionally, univariate and multivariate Cox-regression analyses were performed to identify prognostic factors among patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged over 18 years; (2) Patients with histologically confirmed pancreatic cancer through surgical or puncture procedures; (3) Complete lipid profiles available within one week prior to diagnosis.

Exclusion Criteria:

* (1) Presence of concurrent malignancies; (2) History of previous treatments such as pancreatectomy, chemotherapy, or radiation therapy; (3) Incomplete clinicopathological information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This research involved the inclusion of 364 individuals who were diagnosed with pancreatic cancer at the Affiliated Hospital of Qingdao University from January 2019 to December 2022, following pathological confirmation. The criteria for inclusion were as follows: (1) Adult patients aged over 18 years; (2) Patients with histologically confirmed pancreatic cancer through surgical or puncture procedures; (3) Complete lipid profiles available within one week prior to diagnosis. Exclusion criteria were as follows: (1) Presence of concurrent malignancies; (2) History of previous treatments such as pancreatectomy, chemotherapy, or radiation therapy; (3) Incomplete clinicopathological information.
Sampling Method: Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
OS | 1-30months
  The primary endpoint was overall survival (OS), defined as the time from pathological diagnosis to either death or the most recent follow-up.

SECONDARY OUTCOMES:
PFS | 1-10months
  The secondary measure was the duration from the initial diagnosis to disease progression, referred to as progression-free survival (PFS). Both are measured in months.

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No